CLINICAL TRIAL: NCT00250172
Title: PET Whole Body Biodistribution and Test Retest Brain Imaging Studies Using a Phosphodiesterase 4 Inhibitor (R)-[11C]Rolipram
Brief Title: PET Whole Body Biodistribution and Test Retest Bain Imaging Studies Using a Phosphodiesterase 4 Inhibitor (R)-[11C]Rolipram
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060002; 06-M-0002
Record Dates: First submitted 2005-11-05; First posted 2005-11-07 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-09-15

CONDITIONS: Dosimetry; Healthy
Keywords: Dosimetry; Pharmacokinetics; Compartment Analysis; Reproducibility; Healthy Volunteer; HV

INTERVENTIONS:
Drug: [C-11](R)-rolipram

SUMMARY:
The purpose of this study is to measure a particular protein in the brain called the phosphodiesterase by using the imaging techniques of positron emission tomography (PET) and magnetic resonance imaging (MRI).

...

DETAILED DESCRIPTION:
Both basic and clinical studies have indicated that the 3', 5'-cyclic adenosine monophosphate (cAMP) system plays critical roles in several brain diseases, particularly in mood disorders and drug addiction. cAMP is synthesized from adenosine 5'-triphosphate (ATP) by adenylyl cyclase and metabolized by cyclic nucleotide phosphodiesterases (PDEs). Among components of the cAMP pathway, PDE4 appears to be critical for antidepressant effects. 4-[3-(cyclopentoxyl)-4-methoxyphenyl]-2-pyrrolidone (rolipram) is an inhibitor of PDE4. As a positron emission tomography (PET) brain imaging agent, rolipram has good properties such as high affinity of 1-2 nM and appropriate lipophilicity (Log P) of ~3. A rat study gave an estimation of low radiation absorbed doses of the active enantiomer (R)-[11C]rolipram. ciociWEge quality. Therefore, R-[11C]rolipram is a promising PET ligand. However, radiation absorbed doses have not been estimated from human whole body imaging studies and a method to measure binding of (R)-[11C]rolipram in human brain has not been established.

<TAB>

The purposes of this protocol are to estimate radiation absorbed doses of (R)-[11C]rolipram by performing whole body imaging studies on healthy human subjects and also to establish an accurate method to measure PDE4 levels in brain by performing test retest brain imaging studies. The results of this overall study are required to apply this PET ligand in various neurological and psychiatric disorders in the future.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must be healthy and aged 18 65 years.

EXCLUSION CRITERIA:

PART 1 (WHOLE BODY IMAGING STUDIES):

1. Current psychiatric disease, substance abuse or severe systemic disease based on history and physical exam, poor vision or hearing.
2. Laboratory tests with clinically significant abnormalities.
3. Prior participation in other research protocols or clinical care in the last year such that radiation exposure including that from this protocol would exceed a half of the annual limits. Because human dosimetry of (R)-[(11)C]rolipram has been estimated using rhesus monkeys, the total exposure including that from the (R)-[(11)C]rolipram whole body imaging study will be limited to a half of the RSC guidelines.
4. Pregnancy and breast feeding.
5. Positive HIV test.
6. Positive urine drug screen.

PART 2 (TEST RETEST BRAIN IMAGING STUDIES):

1. Current psychiatric disease, substance abuse or severe systemic disease based on history and physical exam, poor vision or hearing.
2. Laboratory tests with clinically significant abnormalities.
3. Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual limits. Results of part 1 will be used to calculate total radiation exposure within a year.
4. Pregnancy and breast feeding.
5. Claustrophobia.
6. Presence of ferromagnetic metal in the body or heart pacemaker.
7. Positive HIV test.
8. A history of brain disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-10-31; Primary Completion 2009-02-05 (Actual); Study Completion 2009-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Fujita, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abi-Dargham A, Gandelman M, Zoghbi SS, Laruelle M, Baldwin RM, Randall P, Zea-Ponce Y, Charney DS, Hoffer PB, Innis RB. Reproducibility of SPECT measurement of benzodiazepine receptors in human brain with iodine-123-iomazenil. J Nucl Med. 1995 Feb;36(2):167-75. PMID 7830108
- [Background] Cloutier RJ, Smith SA, Watson EE, Snyder WS, Warner GG. Dose to the fetus from radionuclides in the bladder. Health Phys. 1973 Aug;25(2):147-61. doi: 10.1097/00004032-197308000-00009. No abstract available. PMID 4784245
- [Background] Conti M, Nemoz G, Sette C, Vicini E. Recent progress in understanding the hormonal regulation of phosphodiesterases. Endocr Rev. 1995 Jun;16(3):370-89. doi: 10.1210/edrv-16-3-370. No abstract available. PMID 7671852